CLINICAL TRIAL: NCT06385886
Title: Recruitment and Engagement in Care to Impact Practice Enhancement (RECIPE) for Sickle Cell Disease
Acronym: RECIPE
Status: Recruiting | Type: Observational
Sponsor: RTI International (Other)
Responsible Party: Sponsor
Other Study IDs: 1R01HL158807-01A1 (NIH)
Record Dates: First submitted 2023-06-13; First posted 2024-04-26 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease Care; Unaffiliated patients; Linkage Coordinator
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Individuals diagnosed with Sickle Cell Disease (SCD) but not receiving care from an SCD specialist.: Individuals diagnosed with Sickle Cell Disease (SCD) but unaffiliated from SCD specialist care. These individuals will be connected to a linkage coordinator (trained staff) to provide a patient-centered approach to engagement with SCD specialist care.
  Interventions: Behavioral: Linkage Coordinator

INTERVENTIONS:
Behavioral: Linkage Coordinator — The Linkage Coordinator (LC) will be the initial contact with unaffiliated SCD patients to establish a relationship, champion preventative services, and support them in engaging with an SCD specialist by helping patients address barriers to care. Study staff will provide initial and ongoing training to the LC to ensure they have adequate support to effectively engage with patients.

SUMMARY:
The goal of this observational study is to help us understand more about the best ways to help individuals living with Sickle Cell Disease (SCD) get the best care. The main question it aims to answer is: How to find individuals unaffiliated from SCD specialist care use three distinct pathways? Once unaffiliated individuals are found using the pathways, Investigators will employ linkage coordinators (trained staff) to engage these patients in care. Participants will be asked to fill out an assessment survey which will cover areas such as previous and current treatment, clinic and hospital experience, pain, and quality of life. Participants will also be given the option of participation in a 1-hour long interview how they feel about treatment for sickle cell disease including clinic experience, pain, and quality of life?

DETAILED DESCRIPTION:
The goal of RECIPE (Recruitment and Engagement in Care to Impact Practice Enhancement) for Sickle Cell Disease is to find unaffiliated patients with SCD using three distinct pathways (Community, Hospital, Surveillance) engage them in care using linkage coordinators (LCs; a successful method adapted from HIV care), and understand the contextual factors and implementation support needed to ensure these methodologies can be further scaled up at a national level. This study is significant because information about unaffiliated patients with SCD who are not actively engaged in the health system has not been systematically collected and studied in the past. Information comes only from experienced clinicians, community groups, patient advocates, and word of mouth. The lack of data about this population is problematic because current implementation studies focus on the barriers related to affiliated patients, with no known strategies identified to engage unaffiliated patients. No previous studies have evaluated the best methods for locating and then engaging and maintaining unaffiliated patients in specialty SCD care. This study will contribute to the literature by optimizing different pathways for finding unaffiliated patients, as well as providing evidence on what may work best in different clinical care settings and among different patients to address barriers to care in hard-to-reach populations.

ELIGIBILITY:
Inclusion Criteria:

* Persons must be >/= 18 years of age
* Persons must have confirmed SCD
* Persons not seen by a SCD specialist > 1 year +/- 3 months
* Literacy in English will be required of the consenting patient or parent/guardian

Exclusion Criteria:

* Persons < 18 years of age
* Persons that are unable to provide informed consent and do not have a designated care-giver that can consent on his/her behalf
* Persons with sickle cell trait (as per hemoglobin electrophoresis)
* Persons seen by a SCD specialist < 1 year +/1 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with Sickle Celle Disease (SCD) who are unaffiliated from SCD care specialists
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Identification of unaffiliated patients | Beginning of enrollment - end of study (up to 5 years)
  Identification of patients through hospital, surveillance, and community-based pathways.
Affiliation with a Sickle cell disease (SCD)-specific care with SCD specialist | Beginning of enrollment - end of study (up to 5 years)
  Rate of affiliation of participants previously unaffiliated with SCD-specific care with an SCD specialist who are now connected to a linkage coordinator and an SCD-specific care with SCD specialist.

SECONDARY OUTCOMES:
Scale Out to Other SCD Centers - Implementation in at least 2 other SCD Center study sites | After methods are optimized - end of study (up to 5 years)
  Once investigators optimize methods for finding and engaging unaffiliated patients with SCD, it is necessary to expand efforts to other SCD sites. The study will expand to include 2 additional sites and begin to assess rate of affiliation of participants previously unaffiliated with SCD-specific care with an SCD specialist who are now connected to a linkage coordinator and an SCD-specific care with SCD specialist.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Kanter, MD, Principal Investigator — University of Alabama, Birmingham (UAB)
Locations (9):
- United States (9):
  - University of Alabama, Birmingham (UAB), Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of California, San Francisco (UCSF), Oakland, California
  - Augusta University, Augusta, Georgia
  - University of Illinois, Chicago, Illinois
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Tennessee at Memphis, Memphis, Tennessee
  - University of Texas at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided